CLINICAL TRIAL: NCT00351962
Title: Phase I/II Study of Fractionated Stereotactic Radiotherapy for Medically Inoperable Non-Small Cell Lung Cancer (NSCLC) or Metastatic Lung Tumours
Brief Title: Phase I/II Study of Fractionated Stereotactic Radiotherapy for Medically Inoperable NSCLC or Metastatic Lung Tumours
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AHS Cancer Control Alberta (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20131
Record Dates: First submitted 2006-07-11; First posted 2006-07-13 (Estimated); Last update posted 2017-09-21 (Actual); Status verified 2013-07

CONDITIONS: Lung Neoplasms; Lung Cancer
Keywords: lung neoplasms; metastatic lung cancer; stereotactic radiation
MeSH Terms: conditions — Lung Neoplasms

ARMS (2):
- Schedule I (10 fractions) (Experimental): Subjects will receive a total of 10 stereotactic radiation treatments, given over 3 weeks.
  Interventions: Procedure: Fractionated Stereotactic Radiotherapy
- Schedule II (4 fractions) (Experimental): Subjects will receive a total of 4 stereotactic radiation treatments, given over 2 weeks.
  Interventions: Procedure: Fractionated Stereotactic Radiotherapy

INTERVENTIONS:
Procedure: Fractionated Stereotactic Radiotherapy

SUMMARY:
Medically inoperable lung cancer or metastatic lung tumours will be treated with fractionated stereotactic radiation using a schedule of 1) 12 Gy x 4 treatments or 2) 6 Gy x 10 treatments.

DETAILED DESCRIPTION:
You will be positioned in a special body mould while you are lying in the treatment position. This ensures that you are treated in the exact position each time. A soft plastic sheet may be placed over your body from the chest down. A vacuum device may be used to apply the sheet gently over you. This mild compression will ensure that you can breathe comfortably but will minimize any movement which may affect the accuracy of your treatments.

A CT (computed tomography) scan will be done for your treatment planning. The CT scan will take approximately 45 minutes. In some cases, intravenous dye may be administered during the CT scan. You will be asked to hold your breath for a short time during the CT scan. If you are unable to hold your breath comfortably, the scan will be performed during your normal breathing cycle. In some cases, your doctor may also order a PET (positron emission tomography) scan. The treatment planning to be done by your oncologist and physicist will take approximately one to two weeks. After that is completed, your treatments will begin. Each treatment will take about 30 minutes.

If the CT scans show that there is a lot of movement of your lung cancer due to breathing motion, your oncologist may recommend the insertion of a "fiducial" marker to help guide your treatments. An additional consent form will be obtained prior to this procedure. The "fiducial" marker is a tiny gold or stainless steel coil measuring about one inch long. It would be inserted into your lung in or next to the tumour by a respirologist via bronchoscopy under sedation. The procedure would take approximately 30 minutes, and you would be in hospital for about 4 hours. You would meet the respirologist in the clinic in consultation prior to the procedure so that he/she can tell you more about the procedure and assess your case in details to determine if it is safe for you to undergo the procedure. The insertion of the fiducial marker is considered part of your clinical care and a separate consent will be required prior to this procedure. You may choose not to undergo this procedure but still participate in this study. In some cases, your respirologist may have already inserted a fiducial marker at the time of diagnostic bronchoscopy after discussions with yourself and your radiation oncologist. The "fiducial" marker would be used to guide your radiation treatments during your normal breathing cycle.

You will be assigned into one of the two study groups described below depending on the location of your tumour:

Schedule I (10 fractions): You will receive a total of 10 stereotactic radiation treatments, given over 3 weeks.

Schedule II (4 fractions): You will receive a total of 4 stereotactic radiation treatments, given over 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* non-small cell lung cancer less than 6cm; no mediastinal or distant metastases
* Open to Alberta,Canada Residents

Exclusion Criteria:

* tumour size greater than 6cm; inadequate pulmonary function(ie. FEV1 less than 0.8 L), Karnofsky performance status less than 70, multiple co-morbid conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2006-09 (Actual); Primary Completion 2014-07 (Actual); Study Completion 2014-07-02 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity as defined by CTCAE V3 grade 4 or 5. | At the completion of accrual, an analysis with respect to acute toxicity will be performed after all patients have been followed a minimum of 90 days from the start of RT.
  Each schedule will be evaluated according to the occurrence of DLTs observed.

CONTACTS AND LOCATIONS:
Overall Officials: Harold P Lau, MD, Principal Investigator — Tom Baker Cancer Center
Locations (1):
- Tom Baker Cancer Center, Calgary, Alberta, Canada